CLINICAL TRIAL: NCT07281560
Title: ORTHO BRO: Opinions, Perceptions, & Thoughts of British Resident Doctors on Orthopaedics
Brief Title: Opinions, Perceptions, & Thoughts of British Resident Doctors on Orthopaedics
Acronym: ORTHO BRO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25ORT278
Record Dates: First submitted 2025-11-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Perceptions of Orthopaedic Surgery Among UK Resident Doctors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Foundation Doctors: Foundation Year 1 and Year 2 doctors currently employed in the NHS
- Core Trainees: Core Trainees Year 1 and Year 2 currently employed in the NHS
- Non-training/Trust-grade SHOs: Non-training/Trust-grade Senior House Officers currently employed in the NHS

SUMMARY:
Orthopaedic surgery is one of the largest surgical specialties in the UK, delivering high-volume, high-impact care across trauma and elective pathways. Despite this, the specialty continues to face challenges in recruitment, diversity, inclusivity and perceptions of workload and culture. International literature suggests that impressions formed during undergraduate and early postgraduate training strongly influence specialty choice; however, contemporary UK-specific data on how resident doctors view orthopaedics remain limited. The ORTHO BRO Study is a cross-sectional, anonymous online survey designed to capture UK trainees' perceptions of orthopaedics, compare views between those with and without prior orthopaedic rotations, and explore spontaneous associations. Findings will inform training improvement, inclusivity initiatives, and recruitment strategies.

The study targets UK foundation doctors (F1/F2), core trainees (CT1/CT2), and trust-grade/non-training senior house officers (SHOs) across multiple trusts/foundation schools.

ELIGIBILITY:
Inclusion Criteria:

* Are currently employed within the UK National Health Service (NHS) as a Foundation Year 1 (F1), Foundation Year 2 (F2), Core Training Year 1 (CT1), Core Training Year 2 (CT2) or trust-grade/non-training senior house officer (SHO).
* Are aged 18 years or older.
* Are able to read and understand English sufficiently to comprehend the participant information and complete the online questionnaire.
* Are willing and able to provide electronic informed consent before taking part.
* Agree to participate voluntarily and understand that participation is anonymous and non-compulsory.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Foundation Doctors (F1/F2), Core Trainees (CT 1/CT2) and Non-training/Trust-grade senior house officers (SHOs) currently employed in the NHS, regardless of whether they have previously worked or completed a placement in Orthopaedics.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Perceived inclusivity of the specialty | Baseline (At a single time point: at completion of the online survey)
  Measured using responses to: "I would consider orthopaedics to be an inclusive specialty." Quantified on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree).Mean scores will be compared between participants with and without prior orthopaedic experience.
Perceived work-life balance | Baseline (At a single time point: at completion of the online survey)
  Measured using responses to: "I believe orthopaedics offers a good work-life balance." Quantified on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores will be compared between participants with and without prior orthopaedic experience.
Interest in pursuing a career in orthopaedics | Baseline (At a single time point: at completion of the online survey)
  Measured using responses to: "Would you personally consider pursuing a career in orthopaedics?" Quantified on a 5-point Likert scale (definitely no → definitely yes). Used to explore the relationship between perceptions (inclusivity, lifestyle) and career interest.